CLINICAL TRIAL: NCT06046703
Title: Diet Quality of Pregnant Women With a Strict Plant-based Diet Versus an Omnivorous Diet: a Focus on Vitamin B12 Intake and Other Nutritional and Pregnancy-related Outcomes
Brief Title: Diet Quality of Pregnant Women With a Strict Plant-based Diet Versus an Omnivorous Diet
Status: Not yet recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL84796.068.23
Record Dates: First submitted 2023-08-29; First posted 2023-09-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-10

CONDITIONS: Vitamin B 12 Deficiency; Pregnancy; Nutrient Deficiency; Dietary Exposure
Keywords: vegan diet; pregnancy; vitamin b12; omnivorous; nutrition
MeSH Terms: conditions — Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vegan: Pregnant women with a strict plant-based diet
  Interventions: Other: Daily nutritional intake
- Omnivorous: Pregnant women with an omnivorous diet.
  Interventions: Other: Daily nutritional intake

INTERVENTIONS:
Other: Daily nutritional intake — Nutritional intake with a focus on vitamin B12, but also other micronutrients and macronutrients

SUMMARY:
The goal of this observational study is to compare the nutritional intake among pregnant women with a strict plant-based diet versus an omnivorous diet.

The main aim is to compare vitamin B12 intake.

Participants will be asked to:

* fill out a health questionnaire
* fill out a three-day food diary
* undergo blood sampling Researchers will compare pregnant women with a strict plant-based diet and pregnant women with an omnivorous diet to see if their nutritional intake is comparable.

DETAILED DESCRIPTION:
The number of people adhering to a strict plant-based diet is increasing globally. Adequate maternal nutrition during pregnancy is essential for fetal development, as deficiencies in macro- and micronutrients can cause maternal and neonatal complications. Nutrition can play a role in developing pre-eclampsia, premature birth, and intra-uterine growth restriction. Although there is evidence of nutrient deficiencies in people who follow a strict plant-based diet and the significance of maternal diet for both maternal and fetal outcomes, there has been limited research on the nutritional intake and outcomes of pregnant women on a strict plant-based diet. Additionally, to the best of our knowledge, very limited research has been published on the incidence of pregnancy-induced hypertension, pre-eclampsia, gestational diabetes, or pre-term birth in women on a strict plant-based diet. The relation between these outcomes and nutritional intake/status is also unknown in this specific group of women, even though the number of people with a strict plant-based diet is increasing. The only two studies that studied pregnancy-related outcomes in women on a strict plant-based diet were performed in Israel and were not powered to show statistical differences between a strict plant-based diet and obstetrical outcomes. Additionally, the dietary intake in Israel differs from other parts of the world. Thus, it is impossible to ascertain if the results also apply to a population with a distinct diet. Recently, the Royal Dutch Organization of Midwives (Koninklijke Nederlandse Organisatie van Verloskundigen, KNOV) published 'the guide for vegetarian and vegan diet in pregnancy .' They acknowledge the limited availability of scientific research concerning the strict plant-based diet in pregnancy and the non-existence of data on Dutch pregnant women. They recommend performing additional blood tests for vitamin B12 and D in case of possible nutrition deficiencies in this group of pregnant women. A significantly lower ferritin level is also described in pregnant women on a strict plant-based diet. In conclusion, even though the nutritional intake during pregnancy is vital for both mother and child, the nutritional intake amongst Dutch women on a strict plant-based diet during pregnancy is unknown. Previously published results from Israeli women do not apply to the Dutch population, as nutritional intake differs between countries. The recently published KNOV guide suggests checking vitamin blood levels during pregnancy. To advise and update guidelines for Dutch women on a strict plant-based diet during pregnancy, additional research on nutritional intake and the nutritional status of Dutch women on a strict plant-based diet and to compare this with nutritional status of omnivorous pregnant women is crucial.

The participant will complete a health-related questionnaire. The estimated time required to complete the questionnaire is approximately 10 minutes. Additionally, between 27 and 30 weeks of pregnancy, participants will fill out a three-day food diary. It is estimated that the questionnaire will take approximately 30 minutes to complete each day. Finally, the participants must complete a questionnaire following the baby's delivery. This questionnaire will cover various aspects, such as the pregnancy, delivery, and blood results obtained during pregnancy. The estimated time required to complete the questionnaire is approximately 15 minutes.

During the blood sampling, 10 ml of blood will be collected using an evacuated tube system through venepuncture. Taking blood samples is a routine part of clinical practice, not solely for this study. Pregnant women typically undergo venipuncture between 27 and 30 weeks as part of regular obstetrical care.

The study's results will provide valuable information about the nutritional intake and status of pregnant women who follow a strict plant-based diet compared to those who follow an omnivorous diet during pregnancy. It will also examine the impact of these diets on the health of both the mother and fetus. This information can be used in developing and improving guidelines on diet in pregnancy and may contribute to the health of pregnant women and their newborn future children in the future.

ELIGIBILITY:
Inclusion Criteria:

* Before 27 weeks of pregnancy
* Age >18 years
* Strict plant-based diet (vegan diet), defined as a diet without ingestion of animal products (i.e., intake less than once a month during) the entire pregnancy or omnivorous diet, defined as a diet that includes meat
* Willing and able to give written informed consent and to understand, participate and comply with the research project requirements

Exclusion Criteria:

* Food allergy that influences the nutritional intake, e.g., milk allergy, celiac disease, and lactose intolerance
* Medical history of gastrointestinal diseases such as Crohn's disease and other diseases associated with vitamin B12 deficiencies such as (pre-existing) diabetes.
* Medical history of abdominal surgery interfering with nutrient uptake, such as gastric bypass and intestinal resections
* Pre-existing cardio-vascular diseases or auto-immune diseases
* Insufficient understanding of the Dutch language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women from the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 256 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin B12 intake in mcg/day | Participants will fill out the food diary between 27 and 30 weeks of pregnancy
  Participants will fill out a three-day food diary in an app. The vitamin B12 intake will be extracted from this.

SECONDARY OUTCOMES:
Nutritional intake | Participants will fill out the food diary between 27 and 30 weeks of pregnancy
  Participants will fill out a three-day food diary in an app. The intake of micronutrients and macronutrients will be extracted from this app and displayed as a percentage of the daily recommended nutritional intake.
Plasma vitamin B12 | Participants will time the blood draw within 2 weeks after filling out the food diary between 27 en 30 weeks of pregnancy
  Obtaining blood samples from pregnant women for hemoglobin testing is a routine part of clinical practice between 27 and 30 weeks of pregnancy, and not specifically for this study. For study purposes, 10 milliliter (mL) of additional blood will be sampled per participant during this blood withdrawal. Plasma vitamin B12 will be shown in pmol/L.
Plasma vitamin D | Participants will time the blood draw within 2 weeks after filling out the food diary between 27 en 30 weeks of pregnancy
  Obtaining blood samples from pregnant women for hemoglobin testing is a routine part of clinical practice between 27 and 30 weeks of pregnancy, and not specifically for this study. For study purposes, 10mL of additional blood will be sampled per participant during this blood withdrawal. Plasma vitamin D will be shown in nmol/L.
Plasma ferritin | Participants will time the blood draw within 2 weeks after filling out the food diary between 27 en 30 weeks of pregnancy
  Obtaining blood samples from pregnant women for hemoglobin testing is a routine part of clinical practice between 27 and 30 weeks of pregnancy, and not specifically for this study. For study purposes, 10mL of additional blood will be sampled per participant during this blood withdrawal. Plasma ferritin will be shown in µg/L.
Plasma hemoglobin | Participants will time the blood draw within 2 weeks after filling out the food diary between 27 en 30 weeks of pregnancy
  Obtaining blood samples from pregnant women for hemoglobin (mmol/L) testing is a routine part of clinical practice between 27 and 30 weeks of pregnancy, and not specifically for this study.
Maternal and fetal outcomes | Participants will fill in the questionnaire between 6 weeks (min) and 6 months (max) postpartum
  Participants will fill out a questionnaire after the delivery of the baby with questions about: gestational age at delivery, gestational diabetes, pregnancy-induced hypertension, pre-eclampsia, gestational weight gain, birthweight

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Scheepers, Dr., Principal Investigator — Maastricht University Medical Center

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT06046703/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT06046703/ICF_001.pdf